CLINICAL TRIAL: NCT00000732
Title: Evaluation of the Interaction Between Low Dose Trimethoprim/Sulfamethoxazole and Zidovudine
Brief Title: Evaluation of the Interaction Between Low Dose Sulfamethoxazole-Trimethoprim and Zidovudine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 033; 11009 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Drug Interactions; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — HIV Infections; Pneumonia, Pneumocystis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Zidovudine

INTERVENTIONS:
Drug: Sulfamethoxazole-Trimethoprim
Drug: Zidovudine

SUMMARY:
To determine if the pharmacokinetics of low doses of zidovudine (AZT) (that is, how fast AZT reaches the blood, what concentration of AZT is attained in the blood, and how long AZT remains in the blood) changes from day-to-day in the same patient. Also to determine whether the pharmacokinetics of AZT is changed by sulfamethoxazole/trimethoprim (SMX/TMP) given at the same time or whether the pharmacokinetics of SMX/TMP is altered by AZT therapy. AZT has been effective in treating some patients with AIDS, and SMX/TMP is an antibiotic combination which is useful in preventing or treating Pneumocystis carinii pneumonia (PCP), which is an important cause of disease and death in patients with AIDS. It is important to know how drugs interact in patients because addition of a second drug may change the speed at which a drug is eliminated from the body, and cause increased toxic effects or decreased therapeutic effects.

DETAILED DESCRIPTION:
AZT has been effective in treating some patients with AIDS, and SMX/TMP is an antibiotic combination which is useful in preventing or treating Pneumocystis carinii pneumonia (PCP), which is an important cause of disease and death in patients with AIDS. It is important to know how drugs interact in patients because addition of a second drug may change the speed at which a drug is eliminated from the body, and cause increased toxic effects or decreased therapeutic effects.

Patients take AZT every 4 hours and/or SMX/TMP every 12 hours by mouth for 4 days as outpatients and then come into the clinical research center for 2 days of studies. On day 5 the final dose of medicine is given orally (SMX/TMP) or by intravenous infusion (AZT). Blood samples are drawn 10-20 times over a period of 12 hours and urine is collected for 36 hours. Concentrations of the drugs in the blood and urine samples are determined. This sequence is repeated twice, so that each patient takes AZT alone, SMX/TMP alone, and the combination of AZT and SMX/TMP over a period of about 3 weeks. Patients may be included in the study if they are asymptomatic, or have been diagnosed with ARC or AIDS, but not if they have PCP or any other severe opportunistic infection.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Allowed:

* Zidovudine (AZT) for patients with AIDS.
* AIDS related complex (ARC). The presence of any one of the following findings within 12 months prior to entry and the absence of a concurrent illness or conditions other than HIV infection to explain the findings:
* Fever of > 38.5 C degrees persisting for longer than 3 weeks.
* Involuntary weight loss of > 15 lbs. or > 10 percent of baseline noted in a 120-day period prior to evaluation.
* Diarrhea (> 2 liquid stools per day) persisting for longer than 1 month.
* History of clinical diagnosis of oral candidiasis or hairy leukoplakia.
* Patients who have AIDS-defining opportunistic infections or tumors.
* Patients eligible for AZT under the labeling.
* A positive HIV antibody test. Exceptions will be made for patients with a previously positive HIV antibody test with progressive disease and patients where virus isolation has been made.
* A life expectancy of at least 3 months.
* Patient with stable Kaposi's sarcoma, mild herpes infection, mild or stable depression, asymptomatic or mild cytomegalovirus or Epstein-Barr virus infection, or a hepatitis B virus carrier state will be acceptable for study.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Phenytoin.

Prior Medication:

Excluded within 30 days of study entry:

* Other antiretroviral agents.
* Patient has any severe ongoing opportunistic infections including Pneumocystis carinii pneumonia (PCP), cryptococcal or toxoplasmosis meningoencephalitis, disseminated herpes simplex or herpes zoster.
* Patient has significant diarrhea at entry ( > 1 watery stool per day).
* Patient has demonstrated prior sensitivity or has experienced significant adverse effects during prior therapy with the drugs to be used in the study.
* Cannot abstain from alcohol or any other drugs during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Study Completion 1990-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ptachcinski R, Study Chair
Locations (1):
- Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Berson A, Happy K, Rousseau F, Grateau G, Farinotti R, Sereni D. Effect of zidovudine (AZT) on cotrimoxazole (TMP-SMX) kinetics: preliminary results. Int Conf AIDS. 1993 Jun 6-11;9(1):501 (abstract no PO-B30-2193)
- [Background] Canas E, Pachon J, Garcia-Pesquera F, Castillo JR, Viciana P, Cisneros JM, Jimenez-Mejias ME. Absence of effect of trimethoprim-sulfamethoxazole on pharmacokinetics of zidovudine in patients infected with human immunodeficiency virus. Antimicrob Agents Chemother. 1996 Jan;40(1):230-3. doi: 10.1128/AAC.40.1.230. PMID 8787912